CLINICAL TRIAL: NCT03263078
Title: Difference Between Inhalation Anesthesia and Total Intravenous Anesthesia in Free Flap Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: CF16113B
Record Dates: First submitted 2017-08-21; First posted 2017-08-28 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Surgery
Keywords: inhalation,intravenous anesthesia
MeSH Terms: conditions — Respiratory Aspiration | interventions — Propofol; Sevoflurane

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TIVA with Propofol in free flap surgery (Experimental): Total intravenous anesthesia(TIVA) with Propofol
  Interventions: Drug: Propofol
- Sevoflurane in free flap surgery (Active Comparator): Inhalation anesthesia with Sevoflurane
  Interventions: Drug: Sevoflurane

INTERVENTIONS:
Drug: Propofol — For the maintenance of anesthesia, we used 2% propofol (Fresofol®, Fresenius Kabi, Germany) administered by the target controlled infusion (TCI) system (Orchestra® Base Primea; Fresenius Kabi, Germany) in Schnider mode with an effect concentration (Ce) of 2.5-3.5 µg ml-1
  Arms: TIVA with Propofol in free flap surgery
Drug: Sevoflurane — Anesthesia was maintained using 1-3% sevoflurane (ULTANE®, AbbVie Inc., USA) in the Sevoflurane group.
  Arms: Sevoflurane in free flap surgery

SUMMARY:
The purpose of this study is to compare the difference between total intravenous anesthesia to inhaled anesthesia in free flap surgery.

DETAILED DESCRIPTION:
The aim of this study is to perform a randomized controlled trial to examine the effects of different anesthetics on intraoperative hemodynamic stability during free flap surgery and postoperative complications

ELIGIBILITY:
Inclusion criteria:

Patients who need head and neck cancer excision and free flap reconstruction surgery

Exclusion criteria:

1. preoperative cognitive dysfunction, NYHA CHF > III or LVEF < 30%
2. preoperative documented obstructive or restrictive lung disease
3. liver cirrhosis; severe chronic renal insufficiency (GFR < 30 ml·min-1·1.73 m-2.)
4. peripheral arterial occlusive disease expected to be a contraindication for PiCCO catheter insertion
5. Active cardiac arrhythmias that were assumed to preclude valid assessment using arterial pulse contour analysis
6. anticipated bilateral femoral arterial and central venous catheterization when the jugular and subclavian veins were not available due to surgical extent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Number of patients with postoperative pulmonary complication | 1 day
  A radiologist who was unaware of the group assignment evaluated the images and confirmed any PPCs, such as pulmonary edema, pneumonia, pleural effusion or atelectasis

SECONDARY OUTCOMES:
Mean arterial blood pressure, MAP (mmHg) | 1 day
  Measure MAP hourly (T0: First data after monitor instrumentation, T1: first hour, T2: second hour, Tend: at the end of surgery) and compare the difference between groups)
Cardiac index , CI (L·min-1·m-2)) | 1 day
  Measure CI hourly (T0: First data after monitor instrumentation, T1: first hour, T2: second hour, Tend: at the end of surgery) and compare the difference between groups)
Systemic vascular resistance index, SVRI (dynes · sec · cm-5) | 1 day
  Measure SVRI hourly (T0: First data after monitor instrumentation, T1: first hour, T2: second hour, Tend: at the end of surgery) and compare the difference between groups)
Stroke Volume Variation , SVV (%) | 1 day
  Measure SVV hourly (T0: First data after monitor instrumentation, T1: first hour, T2: second hour, Tend: at the end of surgery) and compare the difference between groups)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Chang, MD, Principal Investigator — Anesthesiology Department, Taichung Veterans General Hospital
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwain, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chang YT, Lai CS, Lu CT, Wu CY, Shen CH. Effect of Total Intravenous Anesthesia on Postoperative Pulmonary Complications in Patients Undergoing Microvascular Reconstruction for Head and Neck Cancer: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2022 Sep 15;148(11):1013-21. doi: 10.1001/jamaoto.2022.2552. Online ahead of print. PMID 36107412